CLINICAL TRIAL: NCT05317351
Title: A Prospective Randomized Study Comparing the Adenoma Detection Yield of (i) Standard Colonoscopy ("SC"), (ii) Artificial Intelligence (GI Genius™) ("AI"), and (Iii) Combined Artificial Intelligence (GI Genius™) and G-EYE® Colonoscopy
Brief Title: A Prospective Randomized Study Comparing the Adenoma Detection Yield of SC, AI and Combined AI and G-EYE®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: G-EYE15080
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Colorectal (Colon or Rectal) Cancer; Adenoma
MeSH Terms: conditions — Colonic Neoplasms; Adenoma

STUDY DESIGN:
Intervention Model Description: This is a multicenter, 3-arm, randomized, open-label study. Subjects referred to colonoscopy for screening or surveillance will be randomized in a 2:5:5 into one of the following arms: (i) Standard Colonoscopy, (ii) Artificial Intelligence Aided Colonoscopy (GI Genius™), and (iii) Combined Artificial Intelligence Aided Colonoscopy (GI Genius™) and G-EYE® Balloon Aided Colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Standard Colonoscopy ("SC") (Active Comparator): Subjects enrolled to arm 1 ("SC") will undergo colonoscopy using a standard colonoscope.
  Interventions: Device: Standard Colonoscopy
- Artificial Intelligence Aided Colonoscopy (GI Genius™) ("AI") (Active Comparator): Subjects enrolled to arm 2 ("AI") will undergo colonoscopy using a standard colonoscope aided by Artificial Intelligence (GI Genius™)
  Interventions: Device: Artificial Intelligence Aided Colonoscopy (GI Genius™)
- Combined Artificial Intelligence (GI Genius™) and G-EYE® Colonoscopy (AG) (Experimental): Subjects enrolled to arm 3 ("AG") will undergo colonoscopy using the G-EYE® Colonoscope and Artificial Intelligence Aided Colonoscopy (GI Genius™).
  Interventions: Device: Combined Artificial Intelligence Aided Colonoscopy (GI Genius™) and G-EYE® Balloon Aided Colonoscopy

INTERVENTIONS:
Device: Standard Colonoscopy — Subjects randomized into arm 1 will undergo standard colonoscopy using a standard colonoscope
  Arms: Standard Colonoscopy ("SC")
Device: Artificial Intelligence Aided Colonoscopy (GI Genius™) — Subjects randomized into arm 2 will undergo colonoscopy using a standard colonoscope aided by Artificial Intelligence (GI Genius™)
  Arms: Artificial Intelligence Aided Colonoscopy (GI Genius™) ("AI")
Device: Combined Artificial Intelligence Aided Colonoscopy (GI Genius™) and G-EYE® Balloon Aided Colonoscopy — Subjects enrolled to arm 3 ("AG") will undergo colonoscopy using the G-EYE® Colonoscope and Artificial Intelligence Aided Colonoscopy (GI Genius™).
  Arms: Combined Artificial Intelligence (GI Genius™) and G-EYE® Colonoscopy (AG)

SUMMARY:
This is a multicenter, 3-arm, randomized, open-label study. Subjects referred to colonoscopy for screening or surveillance will be randomized in a 2:5:5 into one of the following arms:

(i) Standard Colonoscopy (ii) Artificial Intelligence Aided Colonoscopy (GI Genius™) (iii) Combined Artificial Intelligence Aided Colonoscopy (GI Genius™) and G-EYE® Balloon Aided Colonoscopy

DETAILED DESCRIPTION:
This is a multicenter, 3-arm, randomized, open-label study. Subjects referred to colonoscopy for screening or surveillance will be randomized in a 2:5:5 into one of the following arms:

(i) Standard Colonoscopy (ii) Artificial Intelligence Aided Colonoscopy (GI Genius™) (iii) Combined Artificial Intelligence Aided Colonoscopy (GI Genius™) and G-EYE® Balloon Aided Colonoscopy Study aim is to compare the adenoma detection yield, expressed by Adenoma Per Colonoscopy (APC), of these 3 arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age ≥ 45 years old
2. Referred to colonoscopy for screening or surveillance colonoscopy (history of adenoma resection)
3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease
2. Subjects with a personal history of polyposis syndrome
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy
4. Subjects with diverticulitis or toxic megacolon
5. Subjects with a history of radiation therapy to abdomen or pelvis
6. Pregnant or lactating female subjects
7. Subjects who are currently enrolled in another clinical investigation.
8. Subjects with current oral or parenteral use of anticoagulants, not considered eligible by the investigator.
9. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
10. Any patient condition deemed too risky for the study by the investigator
11. Previous colonic surgery (except for appendectomy)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2160 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Adenoma Per Colonoscopy (APC) (AI compared with AG) | Upon histology results (up to 30 days)
  Adenoma detection yield, represented by Adenoma Per Colonoscopy (APC) of AI compared with APC of AG.

SECONDARY OUTCOMES:
Adenoma Per Colonoscopy (APC) (SC compared with AG) | Upon histology results (up to 30 days)
  Adenoma detection yield, represented by Adenoma Per Colonoscopy (APC) of SC compared with APC of AG
Advanced Adenoma Per Colonoscopy (AAPC) (SC compared with AG) | Upon histology results (up to 30 days)
  Advanced Adenoma detection yield, represented by Advanced Adenoma Per Colonoscopy (AAPC) of SC compared with AAPC of AG

CONTACTS AND LOCATIONS:
Overall Officials: Douglad K Rex, MD, Principal Investigator — Indina University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: No